CLINICAL TRIAL: NCT04140955
Title: Opioid Tapering After Spine Surgery: a Randomized Controlled Trial
Brief Title: Opioid Tapering After Spine Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, Peter Gaarsdal Uhrbrand, MD, PhD Student, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-16-02-211-19
Record Dates: First submitted 2019-10-22; First posted 2019-10-28 (Actual); Last update posted 2022-10-03 (Actual); Status verified 2022-09

CONDITIONS: Opioid Withdrawal; Postoperative Pain
Keywords: Opioid tapering; Withdrawal symptoms; Spine surgery; Patient satisfaction
MeSH Terms: conditions — Pain, Postoperative; Substance Withdrawal Syndrome; Patient Satisfaction

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tapering plan and telephone counselling (Experimental): Patients receive an individually customized tapering plan at discharge and telephone counselling 5-7 days after discharge.
  Interventions: Procedure: Tapering plan and telephone counselling
- Control group (No Intervention): Patients receive standard care and treatment, i.e. no tapering plan or telephone counselling.

INTERVENTIONS:
Procedure: Tapering plan and telephone counselling — Before discharge, a tapering plan is made in collaboration between the patient and one of the investigators. The telephone counselling will include guidance of the patient and/or adjustments of the tapering plan if needed.
  Arms: Tapering plan and telephone counselling

SUMMARY:
The effect of a tapering plan combined with telephone counselling to assist patients in opioid tapering after surgery remains unexplored. A prospective, randomized controlled trial investigating the effect of a tapering plan in combination with telephone counselling in patients scheduled for spine surgery on a degenerative basis is therefore conducted.

DETAILED DESCRIPTION:
Background with aim:

Preoperative opioid-use is one of the strongest predictors for not tapering off opioids after discharge from surgery. In qualitative studies on chronic opioid use, patients call for further help and assistance in tapering opioids. The aim of this study is to investigate the effect of receiving a tapering plan at discharge and telephone counselling one week after discharge on short and long-term opioid-use in preoperative opioid-users who undergo scheduled spine surgery.

Methods:

One-hundred and ten adult patients scheduled for spine surgery will be included in an investigator-initiated, prospective, randomized, controlled trial with two arms: an intervention arm (receiving tapering plan at discharge and telephone counselling on opioid tapering 5-7 days after discharge) or a control arm (receiving no tapering plan or telephone counselling). The study is approved by the Danish Data Protection Agency (1-16-02-211-19) and the Central Denmark Region Committees on Health Research Ethics (1-10-72-138-19).

Hypothesis:

Our primary hypothesis is that a tapering plan and telephone counselling reduces the percentage of patients who exceed their preoperative opioid consumption from 25% to 5% one month after discharge.

ELIGIBILITY:
Inclusion Criteria:

* Daily opioid consumption at least 14 days before surgery
* Planned degenerative cervical, thoracic or lumbar spine surgery

Exclusion Criteria:

* Severe physical co-morbidity or inability to participate (dementia, language problems or mental illness)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-10-08 (Actual); Study Completion 2020-12-08 (Actual)

PRIMARY OUTCOMES:
Number of patients exceeding their preoperative opioid consumption measured in total Morphine Milligram Equivalents (MME) | 0-30 days after discharge

SECONDARY OUTCOMES:
Number of patients tapering off to zero measured in total MME | 0-90 days after discharge
Withdrawal symptoms (yes/no) during opioid tapering | 0-30 days after discharge
Patient satisfaction (very satisfied, satisfied, neither satisfied nor dissatisfied, dissatisfied, very dissatisfied) | 0-14 days after discharge
Pain-related contacts to the primary and/or secondary health care system (yes/no) | 0-14 days after discharge
Number of patients tapering off to zero measured in total MME | 0-365 days after discharge
Number of patients exceeding their preoperative opioid consumption measured in total Morphine Milligram Equivalents (MME) | 0-365 days after discharge

CONTACTS AND LOCATIONS:
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark

REFERENCES:
- [Derived] Uhrbrand P, Rasmussen MM, Haroutounian S, Nikolajsen L. Shared decision-making approach to taper postoperative opioids in spine surgery patients with preoperative opioid use: a randomized controlled trial. Pain. 2022 May 1;163(5):e634-e641. doi: 10.1097/j.pain.0000000000002456. PMID 34433772
- [Derived] Uhrbrand P, Phillipsen A, Rasmussen MM, Nikolajsen L. Opioid tapering after spine surgery: Protocol for a randomized controlled trial. Acta Anaesthesiol Scand. 2020 Aug;64(7):1021-1024. doi: 10.1111/aas.13576. Epub 2020 Mar 26. PMID 32157678